CLINICAL TRIAL: NCT05002634
Title: Safety of Undenatured Collagen Type II (UCII) Supplement in Healthy Volunteer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Professor, Chulalongkorn University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EC2104220
Record Dates: First submitted 2021-08-03; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Health, Subjective

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- undenatured collagen type II (UCII) supplement (Experimental): The undenatured collagen type II (UCII) supplement 40 mg will be taken once daily for 2 months.
  Interventions: Dietary Supplement: undenatured collagen type II (UCII) supplement

INTERVENTIONS:
Dietary Supplement: undenatured collagen type II (UCII) supplement — The undenatured collagen type II (UCII) supplement 40 mg will be taken once daily for 2 months.
  Other Names: UCII

SUMMARY:
This study will be evaluated safety of undenatured collagen type II (UCII) supplement in 60 healthy volunteer. Liver function test, renal function test, and adverse event will be assessed.

DETAILED DESCRIPTION:
This study will be evaluated safety of undenatured collagen type II (UCII) supplement in 60 healthy volunteer. The undenatured collagen type II (UCII) supplement 40 mg will be taken once daily for 2 months. Liver function test, renal function test, and adverse event will be assessed before and after taking for 1 and 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-60 years
* No taking collagen supplement more than 2 weeks
* No collagen and protein allergy
* No liver and renal disease
* Have a willingness to participate in the study

Exclusion Criteria:

* Uncontrolled disease
* Have complication symptom during study
* Pregnancy or lactation
* Cannot follow the protocol
* During participated in other studies

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-05 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Aspartate aminotransferase value | 2 months
  Aspartate aminotransferase value (U/L) in blood sample

SECONDARY OUTCOMES:
Alkaline phosphatase value | 2 months
  Alkaline phosphatase value (U/L) in blood sample
Alanine transaminase value | 2 months
  Alanine transaminase value(U/L) in blood sample
Blood urea nitrogen value | 2 months
  Blood urea nitrogen value (mg/dl) in blood sample
Creatinine value | 2 months
  Creatinine value (mg/dl) in blood sample
Adverse event | 2 months
  using questionnaire (Yes or No)